CLINICAL TRIAL: NCT04026594
Title: Efficacy of Mindfulness-based Therapy vs. Relaxation in Prevention of Burnout in Medical Students : A Multicenter, Single Blind Randomized Controlled Study
Brief Title: Mindfulness-based Therapy Versus Relaxation in Prevention of Burnout in Medical Students
Acronym: MUSTPrevent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other); University Hospital, Paris (Other); University Hospital, Angers (Other Government); University Hospital, Clermont-Ferrand (Other); University Hospital of Saint-Etienne (Other); University Hospital, Tours (Other); University Hospital, Marseille (Other); University Hospital, Strasbourg (Other); INSERM U1061 Montpellier (Unknown); University Hospital, Toulouse (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RECHMPL19_0063; 2019-A01050-57 (Registry Identifier: ANSM)
Record Dates: First submitted 2019-07-09; First posted 2019-07-19 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Burnout; Emotional Disturbances; Depression
Keywords: burnout prevention; emotional exhaustion; mindfulness; medical students; empathy
MeSH Terms: conditions — Burnout, Psychological; Affective Symptoms; Depression; Emotional Exhaustion | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction (MBSR) (Experimental): 306 participants will be randomized in the MBSR program, consisting of 8 weekly sessions lasting 2 and half hours each. In addition to this, they will be asked to complete 30 minutes of home practice each day. In order to avoid forgetting techniques and to reinforce motivation, a MBSR recall session will be offered six month after intervention.
  All the sessions may be carried out remotely, by videoconference. In this case, both programs should be conducted in this way in order to ensure comparability..
  Interventions: Other: Mindfulness Based Stress Reduction
- Progressive Muscle Relaxation Training (PMRT) (Active Comparator): 306 participants will be randomized in a relaxation program, consisting of 8 weekly sessions lasting 2 and half hours each. In addition to this, they will be asked to complete 30 minutes of home practice each day. In order to avoid forgetting techniques and to reinforce motivation, a relaxation recall session will be offered six month after intervention.
  All the sessions may be carried out remotely, by videoconference. In this case, both programs should be conducted in this way in order to ensure comparability
  Interventions: Other: Relaxation group

INTERVENTIONS:
Other: Mindfulness Based Stress Reduction — MBSR teaches mindfulness meditation and mindful yoga exercises to develop non-judgmental awareness of moment-to-moment experience. The intervention duration is 8 weeks, with weekly two and half hours sessions. It will be delivered according to the fundamental concepts and specific techniques provided in the MBSR manualized protocol by Kabat-Zinn. The program also includes 30-min daily homework exercises.
  MBSR teaches four main mindfulness practices: (1) body scan, a process of moving attention through the body; (2) mindful movement, consisting of gentle yoga stretches to develop awareness of body in movement; (3) sitting meditation; and (4) walking meditation. Inquiry and didactic teaching is also a part of MBSR and allows for some detailed exploration of participants' experiences.
  Arms: Mindfulness Based Stress Reduction (MBSR)
Other: Relaxation group — control group
  Arms: Progressive Muscle Relaxation Training (PMRT)

SUMMARY:
A recent survey exploring mental health in a large cohort of French medical students and young graduates (N = 21.768), observed that 68.2% of participants showed pathologic anxiety. A high level of depressive symptomatology was found in 27.7% of participants, while suicidal ideation was reported by 23.7%. Mindfulness Based Interventions are beneficial for health with a positive impact on mood, anxiety, and well-being. It thus can be hypothesized that such interventions could help to prevent anxio-depressive symptomatology in medical students.

The implementation of prevention programs to promote resilience to stress and empathy among medical students is a priority, included in French National Strategy for Health. Efficacy of Mindfulness Based Interventions in French university must be studied to confirm and strengthen their development. The originality of this project consists in the collaboration of medical schools from different cities and the longitudinal follow-up.

The purpose of this study is to assess the efficacy of a mindfulness-based therapy in burnout prevention in comparison to relaxation.

DETAILED DESCRIPTION:
Recent research highlights the positive impact of Mindfulness-Based Interventions on mental health outcomes and in the development of stress management skills and compassion. Moreover, it has been reported that Mindfulness-Based Interventions are well accepted among university students, mainly because these approaches are seen as emotional skill training rather than a mental health intervention. However, there is a lack of long-term follow-up studies testing the maintenance of benefits.

This study proposes Mindfulness-based interventions for preventive purposes in a large sample of fourth and fifth year medical students from different French cities (Montpellier, Angers, Clermont-Ferrand, Marseille, Nîmes, Paris, Saint-Etienne, Strasbourg, Tours, Lyon and Toulouse) and a one-year follow-up.

The main objective is to assess the efficacy of a Mindfulness Based Stress Reduction (MBSR) (intervention) vs. Progressive Muscle Relaxation Training (PMRT) (control) to prevent burnout (emotional exhaustion) of fourth- and fifth-year medical students after one-year follow-up.

The study also aims to :

1. assess efficacy of MBSR vs. PMRT in fourth- and fifth-year medical students to prevent burnout after six-months (emotional exhaustion, depersonalization and professional achievement) and one year follow-up (depersonalization and professional achievement) ;
2. compare anxio-depressive symptomatology, suicidality, drug consumption, mindfulness skills, empathy, quality of life between pre- and post-intervention, at 6- and 12 months follow-up ;
3. investigate the adherence and acceptability of the protocol ;
4. investigate acceptability and outcomes according to personality traits.

The study is a single blind randomized clinical trial. Overall, 612 students from 11 French universities will be enrolled and assigned randomly to two groups:

1. the MBSR group, which will benefit from a structured 8-week group mindfulness-based stress reduction program;
2. the PMRT group, which will benefit from Progressive Muscle Relaxation Training based on a structured 8-week group program.

Participants will be evaluated at four times: before the intervention (within 8 weeks), within the month following the end of the program, at 6 months and 12 months (+/- 1 month) after the completion of the program. All of the follow-up visits may be carried out remotely. The raters will be blind to treatment allocation (single-blind).

An optional qualitative study will be conducted among 30 students, during the first follow-up visit to assess the subjective experience of participation in relaxation and meditation programs.

The benefits expected from MBSR vs PMRT are to increase mental resources to manage negative emotions and psychological distress, to reduce risk of depression, to increase empathy. The perspectives are to improve the state of the art about the efficacy of MBSR for student's mental health promotion and to help the development of life skills programs for young people and students as proposed by General Direction of Health at the national level. Such programs promote low-cost and safety non-pharmacologic evidence-based interventions for psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled in fourth or fifth year medical study
* Having signed the informed consent
* Being able to attend all scheduled visits and comply with all trial procedures

Exclusion Criteria:

* Suffering from a current depressive episode according to DSM-5 criteria
* Suffering from a current panic disorder according to DSM-5 criteria
* Pregnancy
* Exclusion period in relation to another protocol
* Not being affiliated to the French National Social Security System
* Having reached 4500 € annual compensation for participation in clinical trials
* Protection by law (guardianship or curatorship)
* Deprivation of liberty (by judicial or administrative decision)
* Planned longer stay outside the region that prevents compliance with the visit plan
* For Paris students : participation in the optional teaching "Pleine conscience et médecine" (organized by Cloé Brami)
* For Tours students : participation in the optional teaching on meditation organized by the faculty of medicine
* For Strasbourg students : participation in the optional teaching on meditation (organized by Pr Bloch)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 612 (Estimated)
Dates: Start 2019-10-04 (Actual); Primary Completion 2024-03-04 (Estimated); Study Completion 2024-09-04 (Estimated)

PRIMARY OUTCOMES:
Emotional exhaustion assessed with the Maslach Burnout Inventory (MBI) | at 12 months
  Evaluation of the emotional exhaustion based on the MBI score. The MBI contains three subscales, one of which assesses emotional exhaustion through 9 items. A score below 17 indicates a low degree of emotional exhaustion, a score between 18 and 29 indicates a moderate degree of emotional exhaustion and a score above 30 indicates a high degree of emotional exhaustion. Higher scores reflect greater experienced burnout.

SECONDARY OUTCOMES:
Emotional exhaustion assessed with the Maslach Burnout Inventory (MBI) | at 6 months
  Description: Evaluation of the emotional exhaustion based on the MBI score. The MBI contains three subscales, one of which assesses emotional exhaustion through 9 items. A score below 17 indicates a low degree of emotional exhaustion, a score between 18 and 29 indicates a moderate degree of emotional exhaustion and a score above 30 indicates a high degree of emotional exhaustion. Higher scores reflect greater experienced burnout.
Depersonalization assessed with the Maslach Burnout Inventory (MBI) | at 6 months
  Evaluation of the emotional exhaustion based on the MBI score. The MBI contains three subscales, one of which assesses depersonalization through 5 items. A score below 5 indicates a low degree of depersonalization, a score between 6 and 11 indicates a moderate degree of depersonalization and a score above 12 indicates a high degree of depersonalization. Higher scores reflect greater experienced burnout.
Depersonalization assessed with the Maslach Burnout Inventory (MBI) | at 12 months
  Evaluation of the emotional exhaustion based on the MBI score. The MBI contains three subscales, one of which assesses depersonalization through 5 items. A score below 5 indicates a low degree of depersonalization, a score between 6 and 11 indicates a moderate degree of depersonalization and a score above 12 indicates a high degree of depersonalization. Higher scores reflect greater experienced burnout.
Professional achievement assessed with the Maslach Burnout Inventory (MBI) | at 6 months
  Evaluation of the emotional exhaustion based on the MBI score. The MBI contains three subscales, one of which assesses personal accomplishment through 8 items. A score below 33 indicates a low degree of personal accomplishment, a score between 34 and 39 indicates a moderate degree of personal accomplishment and a score above 40 indicates a high degree of personal accomplishment. Lower scores reflect greater experienced burnout.
Professional achievement assessed with the Maslach Burnout Inventory (MBI) | at 12 months
  Evaluation of the emotional exhaustion based on the MBI score. The MBI contains three subscales, one of which assesses personal accomplishment through 8 items. A score below 33 indicates a low degree of personal accomplishment, a score between 34 and 39 indicates a moderate degree of personal accomplishment and a score above 40 indicates a high degree of personal accomplishment. Lower scores reflect greater experienced burnout.
Psychotropic and analgesic consumption | at 6 months
  Collection of the name and dosage per month for each molecule
Psychotropic and analgesic consumption | at 12 months
  Collection of the name and dosage per month for each molecule
Tobacco consumption | at 6 months
  Number of cigarettes per day within the month
Tobacco consumption | at 12 months
  Number of cigarettes per day within the month
Alcohol consumption | at 6 months
  Frequency of the alcohol consumption within the month
Alcohol consumption | at 6 months
  Quantity of the alcohol consumption within the month
Alcohol consumption | at 12 months
  Frequency of the alcohol consumption within the month
Alcohol consumption | at 12 months
  Quantity of the alcohol consumption within the month
Alcohol consumption assessed with the Alcohol Use Disorders Identification Test (AUDIT) | at 12 months
  Quantity of alcohol consumed within the month as assessed with the AUDIT. Higher scores reflect high risk drinking
Alcohol consumption assessed with the Alcohol Use Disorders Identification Test (AUDIT) | at 12 months
  Frequency of alcohol consumed within the month as assessed with the AUDIT. Higher scores reflect high risk drinking
Drug consumption | at 6 months
  Collection of the name of consumed substances, frequency of the consumption within the month
Drug consumption | at 6 months
  Collection of the name of consumed substances, quantity of the consumption within the month
Drug consumption | at 12 months
  Collection of the name of consumed substances, frequency of the consumption within the month
Drug consumption | at 12 months
  Collection of the name of consumed substances, quantity of the consumption within the month
Drug consumption assessed with the Drug Abuse Screening Test (DAST) | at 12 months
  Drug consumption based on the DAST score. The total score ranges from 0 to 10. The higher the score the greater the problem related to drug consumption.
Cannabis consumption | at 6 months
  Frequency of the cannabis consumption within the month
Cannabis consumption | at 6 months
  Quantity of the cannabis consumption within the month
Cannabis consumption | at 12 months
  Frequency of the cannabis consumption within the month
Cannabis consumption | at 12 months
  Quantity of the cannabis consumption within the month
Cannabis consumption assessed with the Cannabis Abuse Screening Test (CAST) | at 12 months
  Cannabis consumption based on the CAST score. The total score ranges from 0 to 24. The higher the score the greater the problem related to cannabis consumption.
Anxio-depressive symptomatology assessed with the Montgomery Asberg Depression Rating Scale (MADRS) | at 6 months
  Anxio-depressive symptomatology based on the MADRS score. The total score ranges from 0 to 60. Scores between 0 and 6 indicates no depression, scores between 7 and 19 indicates mild depression, scores between 20 and 34 indicates moderate depression and scores above 34 reflects severe depression.
Anxio-depressive symptomatology assessed with the Montgomery Asberg Depression Rating Scale (MADRS) | at 12 months
  Anxio-depressive symptomatology based on the MADRS score. The total score ranges from 0 to 60. Scores between 0 and 6 indicates no depression, scores between 7 and 19 indicates mild depression, scores between 20 and 34 indicates moderate depression and scores above 34 reflects severe depression.
Anxio-depressive symptomatology assessed with the Hospital Anxiety and Depression Scale (HADS) | at 6 months
  Anxio-depressive symptomatology based on the HADS score. The questionnaire is divided in two subscales, one for anxiety and one for depression. Each subscore ranges from 0 to 21. Scores greater than or equal to 11 on either scale indicate anxious or depressive symptomatology.
Anxio-depressive symptomatology assessed with the Hospital Anxiety and Depression Scale (HADS) | at 12 months
  Anxio-depressive symptomatology based on the HADS score. The questionnaire is divided in two subscales, one for anxiety and one for depression. Each subscore ranges from 0 to 21. Scores greater than or equal to 11 on either scale indicate anxious or depressive symptomatology.
Anxio-depressive symptomatology assessed with the Perceived Stress Scale (PSS) | at 6 months
  Anxio-depressive symptomatology based on the PSS score. The total score ranges from 0 to 40. Higher scores reflect greater stress level.
Anxio-depressive symptomatology assessed with the Perceived Stress Scale (PSS) | at 12 months
  Anxio-depressive symptomatology based on the PSS score. The total score ranges from 0 to 40. Higher scores reflect greater stress level.
Anxio-depressive symptomatology assessed with the Numerical Scale for psychological pain | at 6 months
  Anxio-depressive symptomatology based on the Numerical Scale for psychological pain. The questionnaire is divided in three subscales, one for current psychological pain, one for usual psychological pain within the 15 last days and one for maximal psychological pain within the 15 last days. Each scale ranges from 0 to 10. Higher scores indicate greater psychological pain.
Anxio-depressive symptomatology assessed with the Numerical Scale for psychological pain | at 12 months
  Anxio-depressive symptomatology based on the Numerical Scale for psychological pain. The questionnaire is divided in three subscales, one for current psychological pain, one for usual psychological pain within the 15 last days and one for maximal psychological pain within the 15 last days. Each scale ranges from 0 to 10. Higher scores indicate greater psychological pain.
Suicidality assessed with the Columbia Suicide Severity Rating Scale (C-SSRS) | at 6 months
  Evaluation of suicidality through the C-SSRS. The suicidal ideation severity subscale ranges from 1 to 5 (with higher number indicating more severe ideation). The intensity of ideation subscale includes 5 questions each one ranging from 1 to 5 (with higher number indicating more intense ideation). The suicidal behavior subscale includes 4 yes/no questions. The suicidal behavior lethality subscale inquires about the level of actual or potential medical damage.
Suicidality assessed with the Columbia Suicide Severity Rating Scale (C-SSRS) | at 12 months
  Evaluation of suicidality through the C-SSRS. The suicidal ideation severity subscale ranges from 1 to 5 (with higher number indicating more severe ideation). The intensity of ideation subscale includes 5 questions each one ranging from 1 to 5 (with higher number indicating more intense ideation). The suicidal behavior subscale includes 4 yes/no questions. The suicidal behavior lethality subscale inquires about the level of actual or potential medical damage.
Empathy assessed with the Jefferson Scale of Empathy for students | at 6 months
  Evaluation of empathy based on the Jefferson Scale Empathy score. The total score ranges from 20 to 140. Higher scores reflect higher empathy.
Empathy assessed with the Jefferson Scale of Empathy for students | at 12 months
  Evaluation of empathy based on the Jefferson Scale Empathy score. The total score ranges from 20 to 140. Higher scores reflect higher empathy.
Quality of life assessed with the World Health Organization Quality of Life (WHOQOL) | at 6 months
  Quality of life based on the WHOQOL score. The total score ranges from 0 to 100. Higher scores reflect better health.
Quality of life assessed with the World Health Organization Quality of Life (WHOQOL) | at 12 months
  Quality of life based on the WHOQOL score. The total score ranges from 0 to 100. Higher scores reflect better health.
Mindfulness assessed with the Five Facets Mindfulness Questionnaire (FFMQ) | at 6 months
  Evaluation of mindfulness skills based on the FFMQ score. Higher scores indicate higher levels of mindfulness ability.
Mindfulness assessed with the Five Facets Mindfulness Questionnaire (FFMQ) | at 12 months
  Evaluation of mindfulness skills based on the FFMQ score. Higher scores indicate higher levels of mindfulness ability.
Self- compassion assessed with the Self-Compassion Scale (SCS) | at 6 months
  Evaluation of self-compassion skills based on the SCS score. The total score ranges from 26 to 130. Higher scores indicate higher levels of self-compassion.
Self- compassion assessed with the Self-Compassion Scale (SCS) | at 12 months
  Evaluation of self-compassion skills based on the SCS score. The total score ranges from 26 to 130. Higher scores indicate higher levels of self-compassion.
Program adherence | at 12 months
  Program adherence assessed with the number of attended sessions and the rates of dropout.
Program acceptability | at 12 months
  Program acceptability assessed with frequency of formal & informal practice of mindfulness, numerical rating scale for satisfaction and time spent doing exercises per week.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France

REFERENCES:
- [Derived] Baeza-Velasco C, Genty C, Jaussent I, Benramdane M, Courtet P, Olie E. Study protocol of a multicenter randomized controlled trial of mindfulness-based intervention versus relaxation to reduce emotional exhaustion in medical students in France: the "Must prevent" study. BMC Psychiatry. 2020 Mar 11;20(1):115. doi: 10.1186/s12888-020-02529-9. PMID 32160891